CLINICAL TRIAL: NCT00513214
Title: A Phase 1/2a, Double-blind, Placebo-controlled Study of the Safety and Pharmacokinetics of XOMA 052 in Subjects With Type 2 Diabetes Mellitus
Brief Title: Safety and Pharmacokinetics Study of XOMA 052 in Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: XOMA (US) LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: X052073
Record Dates: First submitted 2007-08-07; First posted 2007-08-08 (Estimated); Last update posted 2011-10-04 (Estimated); Status verified 2011-09

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes; Type 2; Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — gevokizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- XOMA 052 (Active Comparator)
  Interventions: Drug: XOMA 052
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XOMA 052 — * Part 1, Single IV infusion at one of six dose levels (mg/kg).
  * Part 2, Single SC injection at one of three dose levels (mg/kg).
  * Part 3, Three biweekly SC injections at one of two dose levels (mg/kg).
  Arms: XOMA 052
Drug: Placebo — * Part 1, Single IV infusion at one of six dose levels (mg/kg).
  * Part 2, Single SC injection at one of three dose levels (mg/kg).
  * Part 3, Three biweekly SC injections at one of two dose levels (mg/kg).
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and pharmacokinetics (PK) of XOMA 052 in subjects with stable Type 2 Diabetes Mellitus (T2D).

The study is a dose-escalation study designed to evaluate route of administration (intravenous or subcutaneous), doses, and dosing regimens for future studies.

ELIGIBILITY:
Inclusion Criteria:

* American Diabetes Association (ADA) diagnostic criteria for T2D - Fasting blood glucose concentration ≥ 126 mg/dL (≥ 7.0 mmol/L) (must be measured within 35 days prior to Day 0) OR Symptoms of hyperglycemia (e.g., thirst, polyuria, weight loss, visual blurring) AND a casual/random plasma glucose value of ≥ 200 mg/dL (≥ 11.1 mmol/L) (must be measured within 35 days prior to Day 0)
* HbA1c ≥ 7.5% and ≤ 12% (DCCT standard)
* Current T2D of duration > 6 months at Screening
* T2D and other diseases must be stable. Stable disease is defined as disease that is judged stable by the investigator and which did not require a change in medications or dosing level on 4 or more consecutive days or 7 days in total within 35 days prior to Day 0.
* Age ≥ 18 and ≤ 70 at Screening
* Weight ≥ 80 lbs (36.3 kg) and ≤ 325 lbs (147.4 kg)
* BMI ≥ 23 and ≤ 40 kg/m2
* For female subjects of child-bearing age, a negative serum pregnancy test. For subjects with reproductive potential, a willingness to use contraceptive measures adequate to prevent the subject or the subject's partner from becoming pregnant during the study.
* Agree not to change diet and exercise regimen during the trial

Exclusion Criteria:

* Use of the following medications - Anti-inflammatory therapy other than aspirin ≤ 100 mg/day; Immunosuppressive treatment; Beta 2 and non-selective adrenergic blockers (Note: selective beta 1 blockers are permitted); Thiazolidinediones; Glucagon-like peptide (GLP) agonists including DPP4 inhibitors
* Change in medication for diabetes within 35 days prior to Day 0, defined as a change in dosing level on 4 or more consecutive days or 7 days in total
* Fasting C-peptide < 400 pM (< 1.20 μg/L)
* Hemoglobin < 8.0 g/dL, WBC < 3.0 X 103/mm3, platelet count < 125 X 103/mm3, creatinine > 1.5 mg/dL, AST/ALT > 2 X ULN, alkaline phosphatase > 2 X ULN
* Positive for GAD65 or IA-2 auto-antibodies
* Known HIV antibody, hepatitis B surface antigen, and/or hepatitis C antibody
* History of malignancy within 5 years prior to study entry other than carcinoma in situ of the cervix, or adequately treated, non-metastatic squamous or basal cell carcinoma of the skin
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
* History of tuberculosis, positive PPD test, active atopic disease requiring medication, or asthma
* Infectious disease - CRP > 30 mg/L, fever, or infection requiring treatment with antibiotics within 3 weeks prior to Screening; History of recurrent infection or predisposition to infection; Active leg or foot ulcer
* Immunodeficiency
* Female subjects who are pregnant, planning to become pregnant during the course of the study, or breast-feeding
* History or symptoms of a demyelinating disease
* Clinically significant diabetic macular edema and/or proliferative diabetic retinopathy by history or fundoscopy
* Receipt of a live (attenuated) vaccine within 3 months prior to Screening
* Major surgery within 35 days prior to Day 0
* Participation in an investigational drug or device trial within 30 days prior to Screening
* Use of a therapeutic monoclonal antibody within 90 days prior to Screening
* Any condition which, in the opinion of the investigator, would jeopardize the subject's safety following exposure to the study drug

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2007-07; Primary Completion 2009-06 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Safety assessed by pre- and post-treatment serial measurements of vital signs. | Part 1: Day 0 pre-treatment through Day 56. Part 2: Day 0 pre-treatment through Day 56. Part 3: Day 0 pre-treatment through Day 84.
Safety assessed by treatment-emergent adverse events. | Part 1: Day 0 post-treatment through Day 56. Part 2: Day 0 post-treatment through Day 56. Part 3: Day 0 post-treatment through Day 84.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Urquilla, MD, Study Director — XOMA (US) LLC
Locations (4):
- United States (4):
  - Escondido, California
  - Miami Gardens, Florida
  - Omaha, Nebraska
  - San Antonio, Texas